CLINICAL TRIAL: NCT02074514
Title: A Phase 3b, Multi-Center, Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of Sofosbuvir Plus Ribavirin in Treatment-Naïve Adults With Chronic Genotype 1 or 3 Hepatitis C Virus Infection
Brief Title: Safety and Efficacy of Sofosbuvir Plus Ribavirin in Treatment-Naive Adults With Chronic Genotype 1 or 3 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0116
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sofosbuvir+RBV 16 weeks (Experimental): Participants with HCV genotypes 1 and 3 will receive sofosbuvir plus ribavirin for 16 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- Sofosbuvir+RBV 24 weeks (Experimental): Participants with HCV genotypes 1 and 3 will receive sofosbuvir plus ribavirin for 24 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — 200 mg tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study will evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir (SOF) + ribavirin (RBV) in treatment-naive adults with chronic genotype 1 or 3 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA ≥10^4 IU/mL at screening
* Confirmed chronic HCV genotype 1 or 3 infection
* HCV treatment naive
* Approximately 30% of individuals may have compensated cirrhosis at screening

Exclusion Criteria:

* Any other chronic liver disease
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Current or prior history of clinical hepatic de-compensation
* Contraindication to RBV therapy, e.g., history of clinically significant hemoglobinopathy (sickle cell disease, thalassemia).
* Chronic use of systemically administered immunosuppressive agents
* History of solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kersey, MSc, Study Director — Gilead Sciences
Locations (12):
- India (12):
  - Hyderabad, Andhra Pradesh
  - Chandigarh, Chandigarh
  - Surat, Gujarat
  - Gurgaon, Haryana
  - Kochi, Kerala
  - Mumbai, Maharashtra
  - New Delhi, National Capital Territory of Delhi
  - Ludhiana, Punjab
  - Jaipur, Rajasthan
  - Coimbatore, Tamil Nadu
  - Lucknow, Uttar Pradesh
  - Kolkata, West Bengal

REFERENCES:
- [Result] Shah S, Acharya SK, Mehta R., Kapoor D, Duseja A, Koshy A, et al. (2016) "Sofosbuvir Plus Ribavirin in the Treatment of Chronic HCV Infection in India." Hepatol Int. 10 (Suppl 1): S15.
- [Result] Shah S, Chowdhury A, Mehta R, Kapoor D, Duseja A, Koshy A, et al. Sofosbuvir plus Ribavirin Results in High SVR4 Rates in Patients with Chronic HCV Genotype 1 or 3 Infection in India (Poster L-47). 56th Annual Conference of Indian Society of Gastroenterology; 2015, November, 19-22 Indore, India.
- [Derived] Shah SR, Chowdhury A, Mehta R, Kapoor D, Duseja A, Koshy A, Shukla A, Sood A, Madan K, Sud R, Nijhawan S, Pawan R, Prasad M, Kersey K, Jiang D, Svarovskaia E, Doehle B, Kanwar B, Subramanian M, Acharya SK, Sarin S. Sofosbuvir plus ribavirin in treatment-naive patients with chronic hepatitis C virus genotype 1 or 3 infection in India. J Viral Hepat. 2017 May;24(5):371-379. doi: 10.1111/jvh.12654. Epub 2016 Dec 9. PMID 27933698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in India. The first participant was screened on 31 March 2014. The last study visit occurred on 30 November 2015.
Groups:
- SOF+RBV 16 Weeks: Sofosbuvir (Sovaldi®; SOF) 400 mg tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 16 weeks.
- SOF+RBV 24 Weeks: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks.
Period: Overall Study
Arm/Group | SOF+RBV 16 Weeks | SOF+RBV 24 Weeks
Started | 59 | 58
Completed | 56 | 54
Not Completed | 3 | 4
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrew Consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least one dose of study drug.
Groups:
- SOF + RBV 16 Weeks GT1: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 16 weeks in participants with genotype (GT) 1 HCV infection
- SOF + RBV 24 Weeks GT1: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks in participants with genotype 1 HCV infection
- SOF + RBV 16 Weeks GT3: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 16 weeks in participants with genotype 3 HCV infection
- SOF + RBV 24 Weeks GT3: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks in participants with genotype 3 HCV infection
- Total: Total of all reporting groups
Arm/Group | SOF + RBV 16 Weeks GT1 | SOF + RBV 24 Weeks GT1 | SOF + RBV 16 Weeks GT3 | SOF + RBV 24 Weeks GT3 | Total
Number analyzed (Participants) | 30 | 28 | 29 | 30 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (11.7) | 46 (12.6) | 40 (12.7) | 37 (10.8) | 42 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 12 | 5 | 42
  Male | 19 | 14 | 17 | 25 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 30 | 28 | 29 | 30 | 117
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 28 | 24 | 26 | 28 | 106
  Not Permitted | 2 | 4 | 3 | 2 | 11
HCV genotype [Number; unit: participants]
  Genotype 1a | 5 | 5 | 0 | 0 | 10
  Genotype 1b | 25 | 23 | 0 | 0 | 48
  Genotype 3 | 0 | 0 | 29 | 30 | 59
Cirrhosis Status [Number; unit: participants]
  Absence | 20 | 19 | 22 | 23 | 84
  Presence | 10 | 9 | 7 | 7 | 33
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.44) | 5.9 (0.72) | 6.2 (0.68) | 6.5 (0.70) | 6.3 (0.67)
IL28b Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 14 | 15 | 17 | 23 | 69
    CT | 13 | 8 | 11 | 7 | 39
    TT | 3 | 5 | 1 | 0 | 9
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 5 | 14 | 10 | 6 | 35
  ≥ 800,000 IU/mL | 25 | 14 | 19 | 24 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set (FAS): participants with genotype 1 or 3 HCV infection who were randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF + RBV 16 Weeks GT1 | SOF + RBV 24 Weeks GT1 | SOF + RBV 16 Weeks GT3 | SOF + RBV 24 Weeks GT3
Number analyzed (Participants) | 30 | 28 | 29 | 30
percentage of participants | 90 [73.5 to 97.9] | 96.4 [81.7 to 99.9] | 100.0 [88.1 to 100.0] | 93.3 [77.9 to 99.2]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- SOF + RBV 16 Weeks: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 16 weeks
- SOF + RBV 24 Weeks: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks
Arm/Group | SOF + RBV 16 Weeks | SOF + RBV 24 Weeks
Number analyzed (Participants) | 59 | 58
percentage of participants | 0 | 3.4

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF + RBV 16 Weeks GT1 | SOF + RBV 24 Weeks GT1 | SOF + RBV 16 Weeks GT3 | SOF + RBV 24 Weeks GT3
Number analyzed (Participants) | 30 | 28 | 29 | 30
percentage of participants
  SVR4 | 90.0 [73.5 to 97.9] | 96.4 [81.7 to 99.9] | 100.0 [88.1 to 100.0] | 96.7 [82.8 to 99.9]
  SVR24 | 90.0 [73.5 to 97.9] | 96.4 [81.7 to 99.9] | 100.0 [88.1 to 100.0] | 93.3 [77.9 to 99.2]

4. Secondary Outcome: Percentage of Participants With Virologic Failure and Viral Relapse
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF + RBV 16 Weeks GT1 | SOF + RBV 24 Weeks GT1 | SOF + RBV 16 Weeks GT3 | SOF + RBV 24 Weeks GT3
Number analyzed (Participants) | 30 | 28 | 29 | 30
percentage of participants
  Overall Virologic Failure | 10.0 | 3.6 | 0 | 3.3
  Relapse | 10.0 | 3.6 | 0 | 3.3

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF + RBV 16 Weeks | SOF + RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/58
Other Adverse Events (participants affected / at risk) | 32/59 | 27/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF + RBV 16 Weeks (N=59) | SOF + RBV 24 Weeks (N=58)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF + RBV 16 Weeks (N=59) | SOF + RBV 24 Weeks (N=58)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Haemolysis (Blood and lymphatic system disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 16 | 11
Fatigue (General disorders) | 8 | 2
Pain (General disorders) | 5 | 4
Pyrexia (General disorders) | 5 | 4
Nasopharyngitis (Infections and infestations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years